CLINICAL TRIAL: NCT05012410
Title: Efficacy of the WeCareAdvisor: An Online Tool to Help Caregivers Manage Behavioral and Psychological Symptoms in Persons Living With Dementia
Brief Title: WeCareAdvisor Study for Caregivers of People Living With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: University of California, Davis (Other); National Institute on Aging (NIA) (NIH); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2007007999; 1R01AG061116-01 (NIH)
Record Dates: First submitted 2021-08-06; First posted 2021-08-19 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Dementia; Caregiver Burnout; Caregiver Stress Syndrome; Alzheimer Disease; Frontotemporal Dementia; Vascular Dementia; Dementia With Lewy Bodies
Keywords: dementia; caregiver; alzheimer's disease; memory loss
MeSH Terms: conditions — Dementia; Caregiver Burden; Alzheimer Disease; Frontotemporal Dementia; Dementia, Vascular; Lewy Body Disease; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial involving an immediate treatment group (Group A) and a 3-month waitlist control group (Group B). Also, groups will be randomized to different prompting conditions (email only, telephone and email) to remind participants to use the tool.
Who Masked: Outcomes Assessor
Masking Description: Single blind allocation. Study interviewers will be masked to group allocation. Other research personnel (investigator, project manager, interventionist), may become aware of group allocation. Caregivers will be asked not to disclose to interviewers the group to which they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immediate treatment group with High-Intensity Prompts (Experimental): Caregivers will use the WeCareAdvisor tool for six months and receive telephone and email prompts.
  Interventions: Behavioral: Immediate treatment group with High-Intensity Prompts
- Immediate treatment group with Low-Intensity Prompts (Experimental): Caregivers will use the WeCareAdvisor tool for six months and receive email prompts only.
  Interventions: Behavioral: Immediate treatment group with Low-Intensity Prompts
- Waitlist Control after three months with high-Intensity prompts (Experimental): After three months, caregivers will receive WeCareAdvisor and telephone and email prompts.
  Interventions: Behavioral: Waitlist Control after three months with High-Intensity Prompts
- Waitlist Control after three months with Low-Intensity Prompts (Experimental): After three months, caregivers will receive WeCareAdvisor and email prompts only.
  Interventions: Behavioral: Waitlist Control after three months with Low-Intensity Prompts

INTERVENTIONS:
Behavioral: Immediate treatment group with High-Intensity Prompts — Caregivers in the immediate treatment group with high-intensity prompts will use the WeCareAdvisor tool for 6 months. Caregivers will receive telephone and email prompts to use the tool.
  Arms: Immediate treatment group with High-Intensity Prompts
Behavioral: Immediate treatment group with Low-Intensity Prompts — Caregivers in the immediate treatment group with low-intensity prompts will use the WeCareAdvisor tool for 6 months. Caregivers will receive email prompts to use the tool.
  Arms: Immediate treatment group with Low-Intensity Prompts
Behavioral: Waitlist Control after three months with High-Intensity Prompts — After 3 months, caregivers will use the WeCareAdvisor tool for 3 months. Caregivers will receive telephone and email prompts. Once the caregiver receives the WeCareAdvisor tool, they will receive a weekly automated email as well as a weekly telephone call from study staff to prompt them to use the tool.
  Arms: Waitlist Control after three months with high-Intensity prompts
Behavioral: Waitlist Control after three months with Low-Intensity Prompts — After 3 months, caregivers will use the WeCareAdvisor tool for 3 months. Caregivers will receive email prompts.
  Arms: Waitlist Control after three months with Low-Intensity Prompts

SUMMARY:
The WeCareAdvisor is an online tool to help caregivers manage behavioral and psychological symptoms of people living with dementia. The trial will evaluate its efficacy to reduce caregiver distress, improve confidence managing behaviors, as well as reduce occurrences and severity of behavioral and psychological symptoms.

Visit https://wecareadvisorstudy.com/ for more information.

DETAILED DESCRIPTION:
Caregivers enrolled in the study will use the web-based WeCareAdvisor tool for either three or six months, depending upon group allocation (immediate treatment vs. 3-month waitlist). Caregivers will be interviewed at baseline, 1, 3 and 6 months by telephone to evaluate their health and wellbeing. Also, utilization data of the tool will be captured.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as the primary caregiver to the person living with memory loss or dementia;
* has been a primary caregiver for at least 6 months;
* report managing >1 behavioral symptom(s) in the past month;
* has an email account or smartphone (to receive daily tips and reminder messages);
* English speaking;
* has own smartphone, tablet, laptop, or desktop computer and access to Internet;
* If person living with dementia is on an anti-dementia or psychotropic medication, they must be on a stable dose for at least 60 days prior to enrollment.
* If caregiver is on an anti-depression or other psychotropic medication, they must be on a stable does for at least 60 days prior to enrollment
* Lives in the United States or US territory

Exclusion Criteria:

* Caregiver currently involved in another clinical trial of psychosocial or educational interventions for dementia;
* Caregiver has a visual impairment that prohibits interaction with the tool, and/or have a hearing impairment sufficient to prohibit telephone communication;
* Caregiver reports person living with dementia is not responsive to his/her environment (e.g., unable to understand short commands or recognize a person coming in/out of the room);
* Caregiver reports person living with dementia is an active suicide risk
* Caregiver reports person living with dementia is likely to have an imminent placement in a long-term care facility (within 6 months).
* Either caregiver/person living with dementia has a terminal disease with life expectancy < 6 months, is in active treatment for cancer, or has had more than 3 acute medical hospitalizations over the past year.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Short-term Change in Caregiver Distress with Behaviors | 1 Month
  For each of 13 domains of behavioral symptoms endorsed on the Neuropsychiatric Inventory-Clinician version (NPI-C), caregivers rate level of distress with behavior (0=not distressing to 5=extremely upset)
Long-term Change in Caregiver Distress with Behaviors (3-Months) | 3 months
  For each of 13 domains of behavioral symptoms endorsed on the Neuropsychiatric Inventory-Clinician version (NPI-C), caregivers rate level of distress with behavior (0=not distressing to 5=extremely upset)
Short-Term Change in Caregiver Confidence Managing Behavioral and Psychological Symptoms of Dementia | 1 month
  Caregivers will rate their level of confidence in dementia signs and symptom management using the 25-item Caregiver Confidence in Medical Sign/Symptom Management scale. For each of 13 domains of behavioral symptoms endorsed on the Neuropsychiatric Inventory-Clinician version, caregivers rate confidence managing behaviors (0 = low confidence - 10= high confidence)
Long-Term Change in Caregiver Confidence Managing Behavioral and Psychological Symptoms of Dementia | 3 months
  Caregivers will rate their level of confidence in dementia signs and symptom management using the 25-item Caregiver Confidence in Medical Sign/Symptom Management scale. For each of 13 domains of behavioral symptoms endorsed on the Neuropsychiatric Inventory-Clinician version, caregivers rate confidence managing behaviors (0 (low-confidence - 10- high-confidence))
Short-Term Change in Person Living with Dementia- Frequency of Behaviors by Severity | 1 Month
  Neuropsychiatric Inventory-Clinician version (NPI-C) is a well-validated questionnaire measuring frequency (0=none to 4=very frequently) and severity (0=none to 3=marked)
Long-Term Change in Person Living with Dementia- Frequency of Behaviors by Severity | 3 Months
  Neuropsychiatric Inventory- Clinician version (NPI-C) is a well-validated questionnaire measuring frequency (0=none to 4=very frequently) and severity (0=none to 3=marked)

SECONDARY OUTCOMES:
Short-Term Change in Person with Dementia- Level of Functioning | 1 months
  Caregiver Assessment of Function (CAFU), a psychometrically sound scale measuring # of ADLs/ IADLs needing assistance, and dependence level (1=total dependence to 7=total independence)
Long-Term Change in Person with Dementia- Level of Functioning | 3 months
  Caregiver Assessment of Function (CAFU), a psychometrically sound scale measuring # of ADLs/ IADLs needing assistance, and dependence level (1=total dependence to 7=total independence)
Short-Term Change in Caregiver Upset with Level of Functioning of Person with Dementia | 1 months
  Caregiver Assessment of Function (CAFU), a psychometrically sound scale measuring level of upset with ADLs/ IADLs dependence (0=Not at all to 4=Extremely)
Long-Term Change in Caregiver Upset with Level of Functioning of Person with Dementia | 3 months
  Caregiver Assessment of Function (CAFU), a psychometrically sound scale measuring level of upset with ADLs/ IADLs dependence (0=Not at all to 4=Extremely)
Change in Person with Dementia's Medications | 6 months
  Caregivers are asked to retrieve (e.g., Brown bag review) prescription and non-prescription medications of person living with dementia and relay name, frequency, and dosage for each medication to interviewer. The investigators will track information on changes in psychotropic medication use for persons living with dementia (intensifications, reductions, additions/deletions, or 'prn' or as needed use).
Short Term Change in Caregiver Wellbeing | 1 Month
  The investigators will use the 13-item Perceived Change for Better Index which assesses caregiver perceived change (1= gotten worse to 5= improved a lot) in affective wellbeing, somatic, ability to manage daily care. It is sensitive to change and has strong psychometric properties.
Long Term Change in Caregiver Wellbeing | 3 Months
  The investigators will use the 13-item Perceived Change for Better Index which assesses caregiver perceived change (0=gotten worse to 5=improved a lot) in affective wellbeing, somatic, ability to manage daily care. It is sensitive to change and has strong psychometric properties.
Short Term Change in Caregiver- Negative Communications | 1 Month
  The investigators will use six items from various scales that assess frequency of use (1=Never to 5=Always) of negative communications by caregivers with persons with dementia (yelling, threatening, criticizing, withdrawing from patient, using harsh tone and screaming).
Long Term Change in Caregiver- Negative Communications | 3 Month
  The investigators will use six items from various scales that assess frequency of use (1=Never to 5=Always) of negative communications by caregivers with persons with dementia (yelling, threatening, criticizing, withdrawing from patient, using harsh tone and screaming).
Utilization of tool use | Through study completion, up to 6 months.
  Dashboard data indicating number of times using tool, number of times using each section of the tool, amount of time spent and for each section of the tool, number of DICE sessions started and completed.
Short-Term Change in Person Living with Dementia- Frequency of Behaviors | 1 months
  Neuropsychiatric Inventory- Clinician version (NPI-C) is a well-validated questionnaire measuring frequency (0=none to 4=very frequently) of behavioral symptoms.
Long-Term Change in Person Living with Dementia- Frequency of Behaviors | 3 months
  Neuropsychiatric Inventory- Clinician version (NPI-C) is a well-validated questionnaire measuring frequency (0=none to 4=very frequently) of behavioral symptoms.
Short-Term Change in Person Living with Dementia- Severity of Behaviors | 1 months
  Neuropsychiatric Inventory- Clinician version (NPI-C) is a well-validated questionnaire measuring severity (0=none to 3=marked) of behavioral symptoms.
Long-Term Change in Person Living with Dementia- Severity of Behaviors | 3 months
  Neuropsychiatric Inventory- Clinician version (NPI-C) is a well-validated questionnaire measuring severity (0=none to 3=marked) of behavioral symptoms.
Short-Term Change in Person Living with Dementia- Number of Behaviors | 1 months
  Neuropsychiatric Inventory- Clinician version (NPI-C) is a well-validated questionnaire measuring the number of behavioral symptoms of dementia endorsed (1=yes,0=no).
Long-Term Change in Person Living with Dementia- Number of Behaviors | 3 months
  Neuropsychiatric Inventory- Clinician version (NPI-C) is a well-validated questionnaire measuring the number of behavioral symptoms of dementia endorsed (1=yes,0=no).

CONTACTS AND LOCATIONS:
Overall Officials: Laura N Gitlin, PhD, Principal Investigator — Drexel University; Helen C Kales, MD, Principal Investigator — University of California, Davis
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data will be stored after 7 years following completion of study and reporting of main outcomes.

REFERENCES:
- [Background] Gitlin LN, Bouranis N, Kern V, Koeuth S, Marx KA, McClure LA, Lyketsos CG, Kales HC. WeCareAdvisor, an Online Platform to Help Family Caregivers Manage Dementia-Related Behavioral Symptoms: an Efficacy Trial in the Time of COVID-19. J Technol Behav Sci. 2022;7(1):33-44. doi: 10.1007/s41347-021-00204-8. Epub 2021 Mar 25. PMID 33786370
- [Result] Gitlin LN, Kales HC, Marx K, Stanislawski B, Lyketsos C. A randomized trial of a web-based platform to help families manage dementia-related behavioral symptoms: The WeCareAdvisor. Contemp Clin Trials. 2017 Nov;62:27-36. doi: 10.1016/j.cct.2017.08.001. Epub 2017 Aug 9. PMID 28800895
- [Result] Kales HC, Gitlin LN, Stanislawski B, Myra Kim H, Marx K, Turnwald M, Chiang C, Lyketsos CG. Effect of the WeCareAdvisor on family caregiver outcomes in dementia: a pilot randomized controlled trial. BMC Geriatr. 2018 May 10;18(1):113. doi: 10.1186/s12877-018-0801-8. PMID 29747583